CLINICAL TRIAL: NCT00912132
Title: The National Standard for Normal Fetal Growth
Status: Completed | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: 999909152; 09-CH-N152
Record Dates: First submitted 2009-05-30; First posted 2009-06-03 (Estimated); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Pregnancy; Fetal Growth
Keywords: Fetal Growth; Pregnancy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Maternal blood sample (serum, plasma, white blood cells, red blood cells and PAXgene RNA) at enrollment, 1st, 2nd, 4th follow-up visits, and postpartum
  * Cord blood and placenta of offspring of consenting women collected at delivery

GROUPS / COHORTS (2):
- Low risk singleton cohort: Women with singleton gestations were enrolled between 8w0d and 13w6d and followed up to nine months (2009-2013) in this prospective cohort study. A sub-set of women with and without gestational diabetes were followed up to 6 weeks postpartum. Enrollment was based upon a predefined set of criteria including medical/reproductive history and pre-pregnancy body mass index. Women with a body mass index between 19.0-29.9 kg/m2 were in the low-risk cohort.
- Obese cohort: Women with singleton gestations were enrolled between 8w0d and 13w6d and followed up to nine months (2009-2013) in this prospective cohort study. A sub-set of women with and without gestational diabetes were followed up to 6 weeks postpartum. Enrollment was based upon a predefined set of criteria including medical/reproductive history and pre-pregnancy body mass index. Women with a body mass index between 30.0-44.9 kg/m2 were in the obese cohort.

SUMMARY:
Normal fetal growth is a critical component of a healthy pregnancy and the long-term health of the offspring. Pivotal to understanding the dynamics of human fetal growth and to defining normal and abnormal fetal growth is the development of standards for fetal growth. The study's purpose was to establish standards for normal fetal growth and size for gestational age for 4 racial/ethnic groups of pregnant women with the eventual creation of individualized standards for fetal growth and improvements in fetal weight estimation. These data for a contemporary cohort of pregnant women should provide data for clinical management.

DETAILED DESCRIPTION:
Summary and aims:

Normal fetal growth is a critical component of a healthy pregnancy and the long-term health of the offspring. Pivotal to understanding the dynamics of human fetal growth and to defining normal and abnormal fetal growth is the development of standards for fetal anthropometric parameters measured longitudinally throughout gestation, which, in turn, can be used to develop interval velocity curves and customized for genetic and physiological factors. We propose to conduct a multi-center prospective observational study (1) to establish a standard for normal fetal growth (velocity) and size for gestational age in the U.S. population; (2) to create an individualized standard for fetal growth potential; and (3) to improve accuracy of fetal weight estimation.

Eligibility:

• Healthy, low-risk pregnant women (both obese and nonobese) between the ages of 18 and 40 from each of the following four self-identified race/ethnicity backgrounds: African American, Asian, Caucasian, and Hispanic.

Design:

* Observational cohort design where pregnant women are recruited prior to 13 weeks gestation and followed throughout pregnancy and delivery for women having livebirths.
* After a sonogram at enrollment (10-13 weeks), women were randomized to receive sonograms according to one of the following four schedules: schedule A: 16, 24, 30, 34, and 38 weeks; schedule B: 18, 26, 31, 35, and 39 weeks; schedule C: 20, 28, 32, 36, and 40 weeks; schedule D: 22, 29, 33, 37, and 41 weeks.
* An enrollment interview was followed by depression screening, physical activity, anthropometric assessment and ultrasonology screening for measurement of fetal growth, and at each of the 5 subsequent visits.
* Uterine artery and fetal Doppler studies at selected gestational weeks.
* Women were asked to provide blood samples at enrollment and at follow-up visits at 16-22 weeks, 24-29 weeks, and 34-37 weeks of gestation.
* Neonatal anthropometry completed for all infants within 12-24 hours after birth.
* Cord blood, plasma, and placenta samples were collected for a smaller subsample of newborns.
* Post-study evaluations: Women who were diagnosed with gestational diabetes during pregnancy were asked to return for a follow-up visit 6 weeks after delivery.

Enrollment:

Final recruitment included 2,802 women with singleton pregnancies of which 2,334 were healthy, low-risk women with pre-pregnancy body mass indices (BMI) between 19-29.9 kg/m2. The racial/ethnic distribution of participating women were: Caucasians (n=614), African American (n=611), Hispanics (n=649), and Asians (n=460), and reflects natality characteristics of contemporary U.S. births. An additional 468 obese women (BMI 30-44.9 kg/m2) were also recruited.

Quality Control:

The quality of the ultrasound measures was guaranteed by implementation of: (1) a comprehensive quality control protocol for ante hoc training and credentialing of all site sonographers, developed by the sonology center at Columbia University, and (2) a rigorous protocol for post hoc quality control, whereby a random sample of all scans, stratified by clinical site and visit, was re-measured for accuracy and reliability.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Singleton, viable pregnancy
* 8 plus 0 - 13 plus 6 weeks of gestation
* Maternal age 18 - 40 years
* BMI 19.0 -29.9kg/m(2) for low risk group; BMI 30.0 - 45.0kg/m(2) for obese group
* Firm LMP
* LMP-date and ultrasound date match within 5 days for gestation estimates between 8 weeks + 0 days and 10 weeks + 6 days, 6 days for those between 11 weeks + 0 days and 12 weeks + 6 days, and 7 days for estimates between 13 weeks + 0 days and 13 weeks + 6 days
* No confirmed or suspected fetal congenital structural or chromosomal anomalies
* Expect to deliver at one of the participating hospitals
* No previous participation in the NICHD Fetal Growth Study

EXCLUSION CRITERIA:

* Smoked cigarettes or used illicit drugs in the six months
* Used illicit drugs in the past year
* Having at least 1 alcoholic drink per day
* Conception by ovulation stimulation drugs or assisted reproductive technology
* Chronic hypertension or renal disease under medical supervision
* Asthma requiring weekly medication
* Diabetes mellitus
* Thyroid disease under medical supervision
* Autoimmune disorder (rheumatoid arthritis, lupus, antiphospholipid antibody syndrome,scleroderma)
* Hematologic disorders (chronic anemia, sickle cell disease thrombocytopenia coagulation defects, thrombophilia)
* Cancer
* HIV or AIDS
* Epilepsy or seizure on medication or occurrence within 2 years
* Psychiatric disorder (bipolar disorder, depression, anxiety disorder currently requiring medication)
* Current anorexia nervosa or bulimia
* Previous severe preclampsia, eclampsia, HELLP syndrome
* Previous stillbirth or neonatal death
* Previous very preterm birth (less than 34 weeks)
* Previous low birthweight (less than 2,500 g)
* Previous macrosomia (greater than or equal to 4,500 g)

The following criteria apply only to obese women only:

* Chronic hypertension or high blood pressure requiring two or more medications
* Diabetes while not pregnant
* Chronic renal disease under medical supervision
* Autoimmune disease (rheumatoid arthritis, lupus, antiphospholipid antibody syndrome, scleroderma)
* Psychiatric disorder (bipolar disorder, depression, anxiety disorder currently requiring medication)
* Cancer (currently receiving treatment)
* HIV or AIDS

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women with singleton gestations (n=2,802) were enrolled from 12 U.S. clinical centers. Women were enrolled between 8w0d and 13w6d gestation, as measured by last menstrual period dating consistent with obstetrical ultrasonology.
Sampling Method: Non-Probability Sample
Enrollment: 2802 (Actual)
Dates: Start 2009-05-19; Primary Completion 2013-08-25 (Actual); Study Completion 2013-08-25 (Actual)

PRIMARY OUTCOMES:
Establish a standard for normal fetal growth (velocity) and size for gestational age in the U.S. population. | 3 years
  Fetal growth trajectories were created using 2-D ultrasound fetal biometry including biparietal diameter, head circumference, humerus length, abdominal circumference, and femur length using standardized protocols. Estimated fetal weight (EFW) was calculated.
  Fetal growth trajectories were created using linear mixed models with cubic splines for estimating racial/ethnic specific fetal growth curves for size, methods that accounted for the variation across individual fetuses. For EFW and each individual anthropometric parameter, we tested for overall differences in the racial/ethnic-specific curves using a likelihood-ratio test. When the global test was significant (<.05 level), we tested for week-specific differences by race/ethnicity using Wald tests at each week of gestation. These tests were conducted on the estimated curves with and without adjustment for maternal characteristics.
  A fetal growth velocity standard by maternal race/ethnicity was also created.
Create an individualized standard for fetal growth potential.
  Individualized and customized fetal growth models will be created using two- dimensional ultrasound measures. Individualized or customized definitions of small for gestational age or large for gestational age will be compared to the NICHD Fetal Growth Study singleton standard cut-points of 10th and 90th percentiles, respectively, to see if they improve detection of maternal and neonatal health outcomes.
Improve accuracy of fetal weight estimation.
  Since the last ultrasound exam is scheduled at term, it was expected that many women would deliver within 3 days after the last ultrasound exam. A formula (or formulas) to estimate fetal weight will be created using a multiple linear regression to include not only the 2-D and 3-D sonographic measurements but also factors such as maternal height and weight, sex of the fetus, and glucose challenge test result. We will identify a formula that provides the best estimate of fetal weight, and apply that formula to a validation group. If the sample size allows, we will randomly split the whole cohort into two groups: one group for testing and the other for validation. If the statistical power is insufficient for splitting, we will use cross-validation.

SECONDARY OUTCOMES:
Construct an individualized standard for fundal height.
  We will reevaluate the sensitivity and specificity of the current approach to using fundal height to monitor fetal growth. We will produce an individualized standard for fundal height. We will compare the new standard with the current approach with regard to true positive and true negative values.
Collect blood samples for an etiology study of gestational diabetes and a prediction study of fetal growth restriction and/or overgrowth.
  Blood samples were collected at enrollment, visit 1, visit 2 and visit 4.
Collect placental tissues and cord blood in selected cases and controls for studies on the etiology of idiopathic fetal growth restriction.
  Placental tissue and cord blood at delivery were collected in selected IUGR cases and controls. Placental DNA samples were genotyped. DNA methylation and RNA were quantified.
Collect dietary intake data to study the association between nutrition and fetal growth.
  Food frequency questionnaire was collected at enrollment and 24-h dietary recall at visit 1, visit 2, visit 3, and visit 4.

CONTACTS AND LOCATIONS:
Overall Officials: Germaine M Louis, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (11):
- United States (11):
  - University of Alabama, Birmingham, Alabama
  - Fountain Valley Regional Hospital, Fountain Valley, California
  - University of California-Long Beach, Long Beach, California
  - University of California, Irvine Medical Center, Orange, California
  - Christiana Care Health Services, Newark, Delaware
  - Northwestern University, Chicago, Illinois
  - Saint Peters University Hospital, New Brunswick, New Jersey
  - New York Presbyterian Healthcare System, Flushing, New York
  - Columbia University, New York, New York
  - Women and Infants, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: Yes
Pregnancy and postpartum data will be made accessible in documented repositories and electronic archives after completion of the studies' analytical phases.
Time Frame: After completion of the studies' analytical phases.
Access Criteria: The data, along with a set of guidelines for researchers applying for the data, will be posted to a data-sharing site. All requests for data must include a short protocol with a specific research question and a plan for analysis. Before receiving any analytical file, all users must complete a Data Use Agreement form.
URL: http://brads.nichd.nih.gov

REFERENCES:
- [Background] Zhang C, Hediger ML, Albert PS, Grewal J, Sciscione A, Grobman WA, Wing DA, Newman RB, Wapner R, D'Alton ME, Skupski D, Nageotte MP, Ranzini AC, Owen J, Chien EK, Craigo S, Kim S, Grantz KL, Louis GMB. Association of Maternal Obesity With Longitudinal Ultrasonographic Measures of Fetal Growth: Findings From the NICHD Fetal Growth Studies-Singletons. JAMA Pediatr. 2018 Jan 1;172(1):24-31. doi: 10.1001/jamapediatrics.2017.3785. PMID 29131898
- [Background] Grantz KL, Grewal J, Kim S, Grobman WA, Newman RB, Owen J, Sciscione A, Skupski D, Chien EK, Wing DA, Wapner RJ, Ranzini AC, Nageotte MP, Craigo S, Hinkle SN, D'Alton ME, He D, Tekola-Ayele F, Hediger ML, Buck Louis GM, Zhang C, Albert PS. Unified standard for fetal growth: the Eunice Kennedy Shriver National Institute of Child Health and Human Development Fetal Growth Studies. Am J Obstet Gynecol. 2022 Apr;226(4):576-587.e2. doi: 10.1016/j.ajog.2021.12.006. Epub 2021 Dec 11. No abstract available. PMID 34906542
- [Background] Grantz KL, Kim S, Grobman WA, Newman R, Owen J, Skupski D, Grewal J, Chien EK, Wing DA, Wapner RJ, Ranzini AC, Nageotte MP, Hinkle SN, Pugh S, Li H, Fuchs K, Hediger M, Buck Louis GM, Albert PS. Fetal growth velocity: the NICHD fetal growth studies. Am J Obstet Gynecol. 2018 Sep;219(3):285.e1-285.e36. doi: 10.1016/j.ajog.2018.05.016. Epub 2018 May 24. PMID 29803819
- [Result] Buck Louis GM, Grewal J, Albert PS, Sciscione A, Wing DA, Grobman WA, Newman RB, Wapner R, D'Alton ME, Skupski D, Nageotte MP, Ranzini AC, Owen J, Chien EK, Craigo S, Hediger ML, Kim S, Zhang C, Grantz KL. Racial/ethnic standards for fetal growth: the NICHD Fetal Growth Studies. Am J Obstet Gynecol. 2015 Oct;213(4):449.e1-449.e41. doi: 10.1016/j.ajog.2015.08.032. PMID 26410205
- [Result] Hediger ML, Fuchs KM, Grantz KL, Grewal J, Kim S, Gore-Langton RE, Buck Louis GM, D'Alton ME, Albert PS. Ultrasound Quality Assurance for Singletons in the National Institute of Child Health and Human Development Fetal Growth Studies. J Ultrasound Med. 2016 Aug;35(8):1725-33. doi: 10.7863/ultra.15.09087. Epub 2016 Jun 27. PMID 27353072
- [Result] Grewal J, Grantz KL, Zhang C, Sciscione A, Wing DA, Grobman WA, Newman RB, Wapner R, D'Alton ME, Skupski D, Nageotte MP, Ranzini AC, Owen J, Chien EK, Craigo S, Albert PS, Kim S, Hediger ML, Buck Louis GM. Cohort Profile: NICHD Fetal Growth Studies-Singletons and Twins. Int J Epidemiol. 2018 Feb 1;47(1):25-25l. doi: 10.1093/ije/dyx161. No abstract available. PMID 29025016
- [Derived] Guivarch C, Wu J, Lu R, Grewal J, Yu G, Li LJ, Yang J, Pang WW, Wang DD, Weir NL, Chen Z, Tsai MY, Zhang C. Longitudinal plasma amino acids during pregnancy and neonatal anthropometry: findings from the NICHD Fetal Growth Studies-Singleton Cohort. BMC Med. 2025 Jun 9;23(1):343. doi: 10.1186/s12916-025-04146-3. PMID 40484929
- [Derived] Le R, Biedrzycki RJ, Tekola-Ayele F. Maternal obesity and ancestry distance in influencing birth outcomes. Int J Obes (Lond). 2025 Aug;49(8):1532-1542. doi: 10.1038/s41366-025-01783-9. Epub 2025 Apr 12. PMID 40221546
- [Derived] Wagner KA, Chen Z, Hinkle SN, Gleason JL, Lee W, Grobman WA, Owen J, Newman RB, Skupski DW, He D, Sherman S, Gore-Langton RE, Zhang C, Grewal J, Grantz KL. Relationship between gestational weight gain with fetal body composition and organ volumes in the Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) Fetal Dimensional Study: a prospective pregnancy cohort. Am J Clin Nutr. 2025 Feb;121(2):367-375. doi: 10.1016/j.ajcnut.2024.12.007. Epub 2025 Jan 16. PMID 39909708
- [Derived] Li LJ, Lu R, Rawal S, Birukov A, Weir NL, Tsai MY, Wu J, Chen Z, Zhang C. Maternal plasma phospholipid polyunsaturated fatty acids in early pregnancy and thyroid function throughout pregnancy: a longitudinal study. Am J Clin Nutr. 2024 Apr;119(4):1065-1074. doi: 10.1016/j.ajcnut.2024.02.016. Epub 2024 Feb 24. PMID 38408725
- [Derived] Saeed H, Wu J, Tesfaye M, Grantz KL, Tekola-Ayele F. Placental accelerated aging in antenatal depression. Am J Obstet Gynecol MFM. 2024 Jan;6(1):101237. doi: 10.1016/j.ajogmf.2023.101237. Epub 2023 Nov 25. PMID 38012987
- [Derived] Mitro SD, Sundaram R, Buck Louis GM, Peddada S, Chen Z, Kannan K, Gleason JL, Zhang C, Grantz KL. Associations of Pregnancy Per- and Polyfluoroalkyl Substance Concentrations and Uterine Fibroid Changes across Pregnancy: NICHD Fetal Growth Studies - Singletons Cohort. Environ Health Perspect. 2023 May;131(5):57007. doi: 10.1289/EHP11606. Epub 2023 May 24. PMID 37224071
- [Derived] Grantz KL, Hinkle SN, He D, Owen J, Skupski D, Zhang C, Roy A. A new method for customized fetal growth reference percentiles. PLoS One. 2023 Mar 16;18(3):e0282791. doi: 10.1371/journal.pone.0282791. eCollection 2023. PMID 36928064
- [Derived] Mitro SD, Sundaram R, Chen Z, Peddada S, Buck Louis GM, Zhang C, Grewal J, Gleason JL, Sciscione AC, Grantz KL. Leiomyomata, neonatal anthropometry, and pregnancy outcomes in singleton pregnancies. Ann Epidemiol. 2023 Apr;80:43-52. doi: 10.1016/j.annepidem.2023.02.008. Epub 2023 Feb 21. PMID 36822279
- [Derived] Tesfaye M, Wu J, Biedrzycki RJ, Grantz KL, Joseph P, Tekola-Ayele F. Prenatal social support in low-risk pregnancy shapes placental epigenome. BMC Med. 2023 Jan 8;21(1):12. doi: 10.1186/s12916-022-02701-w. PMID 36617561
- [Derived] Ouidir M, Chatterjee S, Wu J, Tekola-Ayele F. Genomic study of maternal lipid traits in early pregnancy concurs with four known adult lipid loci. J Clin Lipidol. 2023 Jan-Feb;17(1):168-180. doi: 10.1016/j.jacl.2022.10.013. Epub 2022 Nov 17. PMID 36443208
- [Derived] Liu X, Chen L, Fei Z, Zhao SK, Zhu Y, Xia T, Dai J, Rahman ML, Wu J, Weir NL, Tsai MY, Zhang C. Physical activity and individual plasma phospholipid SFAs in pregnancy: a longitudinal study in a multiracial/multiethnic cohort in the United States. Am J Clin Nutr. 2022 Dec 19;116(6):1729-1737. doi: 10.1093/ajcn/nqac250. PMID 36373403
- [Derived] Mitro SD, Peddada S, Chen Z, Buck Louis GM, Gleason JL, Zhang C, Grantz KL. Natural history of fibroids in pregnancy: National Institute of Child Health and Human Development Fetal Growth Studies - Singletons cohort. Fertil Steril. 2022 Oct;118(4):656-665. doi: 10.1016/j.fertnstert.2022.06.028. Epub 2022 Aug 16. PMID 35981916
- [Derived] Vafai Y, Yeung E, Roy A, He D, Li M, Hinkle SN, Grobman WA, Newman R, Gleason JL, Tekola-Ayele F, Zhang C, Grantz KL. The association between first-trimester omega-3 fatty acid supplementation and fetal growth trajectories. Am J Obstet Gynecol. 2023 Feb;228(2):224.e1-224.e16. doi: 10.1016/j.ajog.2022.08.007. Epub 2022 Aug 8. PMID 35952840
- [Derived] Yisahak SF, Hinkle SN, Mumford SL, Gleason JL, Grantz KL, Zhang C, Grewal J. Periconceptional and First Trimester Ultraprocessed Food Intake and Maternal Cardiometabolic Outcomes. Diabetes Care. 2022 Sep 1;45(9):2028-2036. doi: 10.2337/dc21-2270. PMID 35852359
- [Derived] Zhao SK, Yeung EH, Ouidir M, Hinkle SN, Grantz KL, Mitro SD, Wu J, Stevens DR, Chatterjee S, Tekola-Ayele F, Zhang C. Recreational physical activity before and during pregnancy and placental DNA methylation-an epigenome-wide association study. Am J Clin Nutr. 2022 Oct 6;116(4):1168-1183. doi: 10.1093/ajcn/nqac111. PMID 35771992
- [Derived] Tekola-Ayele F, Zeng X, Chatterjee S, Ouidir M, Lesseur C, Hao K, Chen J, Tesfaye M, Marsit CJ, Workalemahu T, Wapner R. Placental multi-omics integration identifies candidate functional genes for birthweight. Nat Commun. 2022 May 2;13(1):2384. doi: 10.1038/s41467-022-30007-1. PMID 35501330
- [Derived] Ghosal S, Grantz KL, Chen Z. Estimation of multiple ordered ROC curves using placement values. Stat Methods Med Res. 2022 Aug;31(8):1470-1483. doi: 10.1177/09622802221094940. Epub 2022 Apr 21. PMID 35450477
- [Derived] Chatterjee S, Zeng X, Ouidir M, Tesfaye M, Zhang C, Tekola-Ayele F. Sex-specific placental gene expression signatures of small for gestational age at birth. Placenta. 2022 Apr;121:82-90. doi: 10.1016/j.placenta.2022.03.004. Epub 2022 Mar 12. PMID 35303517
- [Derived] Ouidir M, Zeng X, Chatterjee S, Zhang C, Tekola-Ayele F. Ancestry-Matched and Cross-Ancestry Genetic Risk Scores of Type 2 Diabetes in Pregnant Women and Fetal Growth: A Study in an Ancestrally Diverse Cohort. Diabetes. 2022 Feb 1;71(2):340-349. doi: 10.2337/db21-0655. PMID 34789498
- [Derived] Ouidir M, Chatterjee S, Mendola P, Zhang C, Grantz KL, Tekola-Ayele F. Placental Gene Co-expression Network for Maternal Plasma Lipids Revealed Enrichment of Inflammatory Response Pathways. Front Genet. 2021 Oct 21;12:681095. doi: 10.3389/fgene.2021.681095. eCollection 2021. PMID 34745199
- [Derived] Li L, Zhu Y, Wu J, Hinkle SN, Tobias DK, Ma RCW, Weir NL, Tsai MY, Zhang C. Changes of Plasma Phospholipid Fatty Acids Profiles in Pregnancy in Relation to the Diagnosis and Treatment of Gestational Diabetes Mellitus. Clin Chem. 2021 Nov 26;67(12):1660-1675. doi: 10.1093/clinchem/hvab169. PMID 34632496
- [Derived] Tesfaye M, Chatterjee S, Zeng X, Joseph P, Tekola-Ayele F. Impact of depression and stress on placental DNA methylation in ethnically diverse pregnant women. Epigenomics. 2021 Sep;13(18):1485-1496. doi: 10.2217/epi-2021-0192. Epub 2021 Sep 29. PMID 34585950
- [Derived] McDonald SM, May LE, Hinkle SN, Grantz KL, Zhang C. Maternal Moderate-to-Vigorous Physical Activity before and during Pregnancy and Maternal Glucose Tolerance: Does Timing Matter? Med Sci Sports Exerc. 2021 Dec 1;53(12):2520-2527. doi: 10.1249/MSS.0000000000002730. PMID 34138816
- [Derived] Li M, Grewal J, Hinkle SN, Yisahak SF, Grobman WA, Newman RB, Skupski DW, Chien EK, Wing DA, Grantz KL, Zhang C. Healthy dietary patterns and common pregnancy complications: a prospective and longitudinal study. Am J Clin Nutr. 2021 Sep 1;114(3):1229-1237. doi: 10.1093/ajcn/nqab145. PMID 34075392
- [Derived] Grantz KL, Ortega-Villa AM, Pugh SJ, Bever A, Grobman W, Newman RB, Owen J, Wing DA, Albert PS. Combination of Fundal Height and Ultrasound to Predict Small for Gestational Age at Birth. Am J Perinatol. 2023 Jan;40(2):155-162. doi: 10.1055/s-0041-1728837. Epub 2021 May 3. PMID 33940642
- [Derived] Tekola-Ayele F, Ouidir M, Shrestha D, Workalemahu T, Rahman ML, Mendola P, Grantz KL, Hinkle SN, Wu J, Zhang C. Admixture mapping identifies African and Amerindigenous local ancestry loci associated with fetal growth. Hum Genet. 2021 Jul;140(7):985-997. doi: 10.1007/s00439-021-02265-4. Epub 2021 Feb 15. PMID 33590300
- [Derived] Vafai Y, Yeung EH, Sundaram R, Smarr MM, Gerlanc N, Grobman WA, Skupski D, Chien EK, Hinkle SN, Newman RB, Wing DA, Ranzini AC, Sciscione A, Grewal J, Zhang C, Grantz KL. Racial/Ethnic Differences in Prenatal Supplement and Medication Use in Low-Risk Pregnant Women. Am J Perinatol. 2022 Apr;39(6):623-632. doi: 10.1055/s-0040-1717097. Epub 2020 Oct 8. PMID 33032328
- [Derived] Ouidir M, Zeng X, Workalemahu T, Shrestha D, Grantz KL, Mendola P, Zhang C, Tekola-Ayele F. Early pregnancy dyslipidemia is associated with placental DNA methylation at loci relevant for cardiometabolic diseases. Epigenomics. 2020 Jun;12(11):921-934. doi: 10.2217/epi-2019-0293. Epub 2020 Jul 17. PMID 32677467
- [Derived] Tekola-Ayele F, Zeng X, Ouidir M, Workalemahu T, Zhang C, Delahaye F, Wapner R. DNA methylation loci in placenta associated with birthweight and expression of genes relevant for early development and adult diseases. Clin Epigenetics. 2020 Jun 3;12(1):78. doi: 10.1186/s13148-020-00873-x. PMID 32493484
- [Derived] Tekola-Ayele F, Zhang C, Wu J, Grantz KL, Rahman ML, Shrestha D, Ouidir M, Workalemahu T, Tsai MY. Trans-ethnic meta-analysis of genome-wide association studies identifies maternal ITPR1 as a novel locus influencing fetal growth during sensitive periods in pregnancy. PLoS Genet. 2020 May 14;16(5):e1008747. doi: 10.1371/journal.pgen.1008747. eCollection 2020 May. PMID 32407400
- [Derived] Li M, Hinkle SN, Grantz KL, Kim S, Grewal J, Grobman WA, Skupski DW, Newman RB, Chien EK, Sciscione A, Zork N, Wing DA, Nageotte M, Tekola-Ayele F, Louis GMB, Albert PS, Zhang C. Glycaemic status during pregnancy and longitudinal measures of fetal growth in a multi-racial US population: a prospective cohort study. Lancet Diabetes Endocrinol. 2020 Apr;8(4):292-300. doi: 10.1016/S2213-8587(20)30024-3. Epub 2020 Mar 2. PMID 32135135
- [Derived] Workalemahu T, Ouidir M, Shrestha D, Wu J, Grantz KL, Tekola-Ayele F. Differential DNA Methylation in Placenta Associated With Maternal Blood Pressure During Pregnancy. Hypertension. 2020 Apr;75(4):1117-1124. doi: 10.1161/HYPERTENSIONAHA.119.14509. Epub 2020 Feb 10. PMID 32078381
- [Derived] Smarr MM, Bible J, Gerlanc N, Buck Louis GM, Bever A, Grantz KL. Comparison of fetal growth by maternal prenatal acetaminophen use. Pediatr Res. 2019 Aug;86(2):261-268. doi: 10.1038/s41390-019-0379-7. Epub 2019 Mar 25. PMID 30911064
- [Derived] Rawal S, Tsai MY, Hinkle SN, Zhu Y, Bao W, Lin Y, Panuganti P, Albert PS, Ma RCW, Zhang C. A Longitudinal Study of Thyroid Markers Across Pregnancy and the Risk of Gestational Diabetes. J Clin Endocrinol Metab. 2018 Jul 1;103(7):2447-2456. doi: 10.1210/jc.2017-02442. PMID 29889229
- [Derived] Zhu Y, Tsai MY, Sun Q, Hinkle SN, Rawal S, Mendola P, Ferrara A, Albert PS, Zhang C. A prospective and longitudinal study of plasma phospholipid saturated fatty acid profile in relation to cardiometabolic biomarkers and the risk of gestational diabetes. Am J Clin Nutr. 2018 Jun 1;107(6):1017-1026. doi: 10.1093/ajcn/nqy051. PMID 29868913
- [Derived] Bever AM, Pugh SJ, Kim S, Newman RB, Grobman WA, Chien EK, Wing DA, Li H, Albert PS, Grantz KL. Fetal Growth Patterns in Pregnancies With First-Trimester Bleeding. Obstet Gynecol. 2018 Jun;131(6):1021-1030. doi: 10.1097/AOG.0000000000002616. PMID 29742672
- [Derived] Grantz KL, Hediger ML, Liu D, Buck Louis GM. Fetal growth standards: the NICHD fetal growth study approach in context with INTERGROWTH-21st and the World Health Organization Multicentre Growth Reference Study. Am J Obstet Gynecol. 2018 Feb;218(2S):S641-S655.e28. doi: 10.1016/j.ajog.2017.11.593. Epub 2017 Dec 22. PMID 29275821